CLINICAL TRIAL: NCT03863080
Title: A Phase 2a, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study With an Open-Label Extension of RVT-1401 in Myasthenia Gravis Patients
Brief Title: A Study of RVT-1401 in Myasthenia Gravis (MG) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT-1401-2002
Record Dates: First submitted 2019-02-20; First posted 2019-03-05 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Myasthenia Gravis
Keywords: IMVT-1401
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Study with an Open-Label Extension
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Regimen A (Experimental): RVT-1401 680 mg weekly for 6 weeks + optional open-label extension (RVT-1401, 340 mg every 2 weeks for 6 weeks)
  Interventions: Drug: RVT-1401
- Regimen B (Experimental): RVT-1401 340 mg weekly for 6 weeks + optional open-label extension (RVT-1401, 340 mg every 2 weeks for 6 weeks)
  Interventions: Drug: RVT-1401
- Placebo (Placebo Comparator): Placebo for 6 weeks + optional open-label extension (RVT-1401, 340 mg every 2 weeks for 6 weeks)
  Interventions: Drug: RVT-1401; Drug: Placebo

INTERVENTIONS:
Drug: RVT-1401 — Subcutaneous administration of RVT-1401
Drug: Placebo — Subcutaneous administration of Placebo
  Arms: Placebo

SUMMARY:
The purpose of the current study is to assess safety/tolerability and key pharmacodynamic (PD) effects that are considered to be associated with clinical benefit (reduction of total IgG and anti-AChR-IgG) in Myasthenia Gravis patients following treatment with RVT-1401 (also known as IMVT-1401) compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. Myasthenia Gravis Foundation of America (MGFA) Class II-IVa and likely not in need of a respirator for the duration of the study as judged by the Investigator.
3. QMG score ≥12 at Screening and Baseline.

Other, more specific inclusion criteria are defined in the protocol.

Exclusion Criteria:

1. Use of rituximab, belimumab, eculizumab or any monoclonal antibody for immunomodulation within 6 months prior to first dosing.
2. Immunoglobulins given by SC, IV (IVIG), or intramuscular route, or plasmapheresis/plasma exchange (PE) within 4 weeks before Screening.
3. Thymectomy performed < 12 months prior to screening.
4. Total IgG level <6 g/L (at screening).
5. Absolute neutrophil count <1500 cells/mm3(at screening).

Other, more specific exclusion criteria are defined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (15):
  - IMC/Diagnostic and Medical Clinic, Mobile, Alabama
  - Phoenix Neurological Associates, Phoenix, Arizona
  - The Neurology Center of Southern California, Carlsbad, California
  - UC Irvine - MDA ALS and Neuromuscular Center, Orange, California
  - Care Access Research, Pasadena, California
  - CSNA, Colorado Springs, Colorado
  - Yale School of Medicine Department of Neurology, New Haven, Connecticut
  - Neurological Services of Orlando, Orlando, Florida
  - Rare Disease Research, Atlanta, Georgia
  - University of Minnesota - Department of Neurology, Minneapolis, Minnesota
  - Dent Institute, Amherst, New York
  - University of Buffalo, Buffalo, New York
  - Hospital for Special Surgery, New York, New York
  - Allegheny Neurological Associates, Pittsburgh, Pennsylvania
  - UTSW James W. Aston Ambulatory Care Center - Neurology Clinic, Dallas, Texas
- Canada (5):
  - University of Alberta Hospitals - Division of Pulmonary Medicine, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network Toronto General Hospital, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 2a, randomized, double-blind (DB), placebo-controlled study with an Open-Label Extension (OLE) that was designed to investigate the safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy of RVT-1401 versus placebo in acetylcholine receptor (AChR) antibody positive myasthenia gravis (MG) participants.
Pre-assignment Details: A total of 17 participants were enrolled in the study. One participant completed the DB period and did not enter the OLE; this participant completed the 12-week post Double-blind Treatment Follow-up Period.
Groups:
- Double-blind Treatment Period: Placebo: Participants were randomized to receive Placebo during the 6-week double blind period. Participants who completed DB Treatment period entered an OLE where they received 340 mg RVT-1401 every 2 weeks (Q2W),x 3 doses followed by a 6-week follow-up period where the participant did not receive any study treatment.
- Double-blind Treatment Period: RVT-1401 340 mg/Week: Participants were randomized to receive 340 mg/week during the 6-week double blind period. Participants who completed DB Treatment period entered an OLE where they received 340 mg RVT-1401 Q2W x 3 doses, followed by a 6-week follow-up period where the participant did not receive any study treatment.
- Double-blind Treatment Period: RVT-1401 680 mg/Week: Participants were randomized to receive 680 mg/week during the 6-week double blind period. Participants who completed DB Treatment period entered an OLE where they received 340 mg RVT-1401 Q2W x 3 doses, followed by a 6-week follow-up period where the participant did not receive any study treatment.
- Open-label Extension Period: RVT-1401 340 mg Biweekly: Participants who completed DB Treatment period entered an OLE where they received 340 mg RVT-1401 Q2W x 3 doses, followed by a 6-week follow-up period where the participant did not receive any study treatment.
Period: Double-Blind Treatment Period (6 Weeks)
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week | Open-label Extension Period: RVT-1401 340 mg Biweekly
Started | 6 | 5 | 6 | 0
Completed | 6 | 5 | 5 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Open Label Extension Period (12 Weeks)
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week | Open-label Extension Period: RVT-1401 340 mg Biweekly
Started | 0 | 0 | 0 | 15
Completed | 0 | 0 | 0 | 9
Not Completed | 0 | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF) comprised of all participants who received at least 1 dose of study medication.
Groups:
- Double-blind Treatment Period: Placebo: Participants were randomized to receive Placebo during the 6-week double blind period. Participants who completed DB Treatment period entered an OLE where they received 340 mg RVT-1401 every 2 weeks (Q2W) x 3 doses, followed by a 6-week follow-up period where the participant did not receive any study treatment.
- Double-blind Treatment Period: RVT-1401 340 mg/Week: Participants were randomized to receive 340 mg/week during the 6-week double blind period. Participants who completed DB Treatment period entered an OLE where they received 340 mg RVT-1401 Q2W x 3 doses, followed by a 6-week follow-up period where the participant did not receive any study treatment. Participants
- Total: Total of all reporting groups
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week | Total
Number analyzed (Participants) | 6 | 5 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.0 (15.40) | 56.8 (22.17) | 70.8 (14.22) | 56.2 (20.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 1 | 7
  Male | 2 | 3 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 5 | 16
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 5 | 6 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Double-Blind Treatment Period: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. SAEs were defined as any untoward medical occurrence that, at any dose: resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event that may have jeopardized the participant or may have required medical or surgical intervention to prevent one of the other outcomes listed in the definition.
Time Frame: Up to Week 18
Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 6 | 5 | 6
Participants
  Any AE | 5 | 4 | 5
  Any SAE | 0 | 0 | 1

2. Primary Outcome: Open-Label Extension Period: Number of Participants Reporting AEs and SAEs
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. TEAEs are defined as those AEs that started or worsened in severity after the initiation of study drug administration. SAEs were defined as any untoward medical occurrence that, at any dose: resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event that may have jeopardized the participant or may have required medical or surgical intervention to prevent one of the other outcomes listed in the definition.
Time Frame: Up to Week 18
Population: Open-label Extension (OLE) Analysis Set comprised of all participants who enrolled in the OLE study phase and received at least 1 dose of study medication in the OLE. Participants were analyzed based on the randomization schedule, regardless of the treatment actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Open-Label Extension Period: RVT-1401 340 mg Biweekly: Participants who completed DB Treatment period entered an OLE where they received 340 mg RVT-1401 every 2 weeks (Q2W) x 3 doses, followed by a 6-week follow-up period where the participant did not receive any study treatment.
Arm/Group | Open-Label Extension Period: RVT-1401 340 mg Biweekly
Number analyzed (Participants) | 15
Participants
  Any AE | 10
  Any SAE | 1

3. Primary Outcome: Double-Blind Treatment Period: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP), pulse rate and temperature were measured after resting for at least 5 minutes in a semi-supine position.
Time Frame: Up to Week 7
Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 6 | 5 | 6
Participants | 0 | 0 | 0

4. Primary Outcome: Open-label Extension Period: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs including SBP, DBP, pulse rate and temperature were measured after resting for at least 5 minutes in a semi-supine position.
Time Frame: Up to Week 18
Population: OLE Analysis Set. Participants were analyzed based on the randomization schedule, regardless of the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 6 | 5 | 4
Participants | 0 | 0 | 0

5. Primary Outcome: Double-blind Treatment Period: Number of Participants With Clinically Significant Changes in Clinical Laboratory Parameters
Description: Clinical laboratory parameters included clinical chemistry, hematology and urinalysis.
Time Frame: Up to Week 7
Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 6 | 5 | 6
Participants | 0 | 0 | 0

6. Primary Outcome: Open-label Extension Period: Number of Participants With Clinically Significant Changes in Clinical Laboratory Parameters
Description: Clinical laboratory parameters included clinical chemistry, hematology and urinalysis.
Time Frame: Up to Week 18
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 6 | 5 | 4
Participants | 0 | 0 | 0

7. Primary Outcome: Double-Blind Treatment Period: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG)
Description: Twelve-lead ECG was performed after 5 minutes of rest in the supine position.
Time Frame: Up to Week 7
Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 6 | 5 | 6
Participants | 0 | 0 | 0

8. Primary Outcome: Open-label Extension Period: Number of Participants With Clinically Significant Changes in ECG
Description: Twelve-lead ECG was performed after 5 minutes of rest in the supine position.
Time Frame: Up to Week 18
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 6 | 5 | 4
Participants | 0 | 0 | 0

9. Primary Outcome: Double-blind Treatment Period: Percent Change From Baseline in Levels of Total Immunoglobulin G (IgG)
Description: Serum samples were collected for the analysis of total immunoglobulin G. Percent change from Baseline was calculated as the mean value at the specified time frame (Week 7) minus the Baseline value, divided by the Baseline value x 100.
Time Frame: Baseline (Day 1) and Up to Week 7
Population: Full Analysis Set comprised of all randomized participants who received at least 1 dose of randomized study medication with at least 1 valid post-treatment value. Only those participants with data available at specified time points has been presented.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 5 | 5 | 5
Percent change | -3.17 (2.97) | -59.49 (3.15) | -77.66 (2.92)
Statistical Analysis 1: Comparison: Double-blind Treatment Period: Placebo vs Double-blind Treatment Period: RVT-1401 340 mg/Week; Test type: Superiority; p < 0.0001, ANCOVA; Least square mean difference = -56.33 — Treatment comparison between Placebo and RVT-1401 340 mg/week of Total IgG levels has been presented
Statistical Analysis 2: Comparison: Double-blind Treatment Period: Placebo vs Double-blind Treatment Period: RVT-1401 680 mg/Week; Test type: Superiority; p < 0.0001, ANCOVA; Least square mean difference = -74.49 — Treatment comparison between Placebo and RVT-1401 680 mg/week of Total IgG levels has been presented

10. Primary Outcome: Double-blind Treatment Period: Percent Change From Baseline in IgG Subclasses 1, 2, 3 and 4
Description: Serum samples were collected for the analysis of IgG 1, 2, 3 and 4 levels. Percent change from Baseline was calculated as the mean value at the specified time frame (Week 7) minus the Baseline value, divided by the Baseline value x 100.
Time Frame: Baseline (Day 1) and Up to Week 7
Population: Full Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 5 | 5 | 4
Percent change
  IgG1 | -3.3 (3.67) | -65.9 (4.02) | -76.3 (3.98)
  IgG2 | -2.2 (5.35) | -54.7 (5.65) | -63.6 (5.60)
  IgG3 | -2.1 (4.69) | -68.2 (5.05) | -82.9 (5.12)
  IgG4 | -3.1 (5.68) | -48.0 (6.08) | -64.7 (6.10)
Statistical Analysis 1: Comparison: Double-blind Treatment Period: Placebo vs Double-blind Treatment Period: RVT-1401 340 mg/Week; Test type: Superiority; p < 0.001, ANCOVA; Least square mean difference = -62.7 — Treatment comparison between Placebo and RVT-1401 340 mg/week of IgG 1 subclass has been presented
Statistical Analysis 2: Comparison: Double-blind Treatment Period: Placebo vs Double-blind Treatment Period: RVT-1401 680 mg/Week; Test type: Superiority; p < 0.001, ANCOVA; Least square mean difference = -73.0 — Treatment comparison between Placebo and RVT-1401 680 mg/week of IgG 1 subclass has been presented
Statistical Analysis 3: Comparison: Double-blind Treatment Period: Placebo vs Double-blind Treatment Period: RVT-1401 340 mg/Week; Test type: Superiority; p < 0.001, ANCOVA; Least square mean difference = -52.5 — Treatment comparison between Placebo and RVT-1401 340 mg/week of IgG 2 subclass has been presented
Statistical Analysis 4: Comparison: Double-blind Treatment Period: Placebo vs Double-blind Treatment Period: RVT-1401 680 mg/Week; Test type: Superiority; p < 0.001, ANCOVA; Least square mean difference = -61.4 — Treatment comparison between Placebo and RVT-1401 680 mg/week of IgG 2 subclass has been presented
Statistical Analysis 5: Comparison: Double-blind Treatment Period: Placebo vs Double-blind Treatment Period: RVT-1401 340 mg/Week; Test type: Superiority; p < 0.001, ANCOVA; Least square mean difference = -66.1 — Treatment comparison between Placebo and RVT-1401 340 mg/week of IgG 3 subclass has been presented
Statistical Analysis 6: Comparison: Double-blind Treatment Period: Placebo vs Double-blind Treatment Period: RVT-1401 680 mg/Week; Test type: Superiority; p < 0.001, ANCOVA; Least square mean difference = -80.8 — Treatment comparison between Placebo and RVT-1401 680 mg/week of IgG 3 subclass has been presented
Statistical Analysis 7: Comparison: Double-blind Treatment Period: Placebo vs Double-blind Treatment Period: RVT-1401 340 mg/Week; Test type: Superiority; p < 0.001, ANCOVA; Least square mean difference = -44.9 — Treatment comparison between Placebo and RVT-1401 340 mg/week of IgG 4 subclass has been presented
Statistical Analysis 8: Comparison: Double-blind Treatment Period: Placebo vs Double-blind Treatment Period: RVT-1401 680 mg/Week; Test type: Superiority; p < 0.001, ANCOVA; Least square mean difference = -61.6 — Treatment comparison between Placebo and RVT-1401 680 mg/week of IgG 4 subclass has been presented

11. Primary Outcome: Double-Blind Treatment Period: Percent Change From Baseline in Anti-acetylcholine Receptor Immunoglobulin G (Anti-AChR-IgG) at Week 7
Description: Serum samples were collected for the analysis of Anti-AChR-IgG. Percent change from Baseline was calculated as the mean value at the specified time frame (Week 7) minus the Baseline value, divided by the Baseline value x 100.
Time Frame: Baseline (Day 1) and Week 7
Population: Full Analysis Set. Only those participants with data available at definite timepoints has been presented.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- Double-blind Treatment Period: RVT-1401 340 mg/Week: Participants were randomized to receive 340 mg/week during the 6-week double blind period. Participants who completed DB Treatment period entered an OLE where they received an additional 3 doses of 340 mg RVT-1401 Q2W x 3 doses, followed by a 6-week follow-up period where the participant did not receive any study treatment.
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 5 | 5 | 4
Percent change | 15.92 (12.41) | -46.66 (13.64) | -85.28 (12.27)
Statistical Analysis 1: Comparison: Double-blind Treatment Period: Placebo vs Double-blind Treatment Period: RVT-1401 340 mg/Week; Test type: Superiority; p = 0.0009, ANCOVA; Least square mean difference = -62.58 — Treatment comparison between Placebo and RVT-1401 340 mg/week of Anti-AChR-IgG has been presented
Statistical Analysis 2: Comparison: Double-blind Treatment Period: Placebo vs Double-blind Treatment Period: RVT-1401 680 mg/Week; Test type: Superiority; p < 0.0001, ANCOVA; Least square mean difference = -101.20 — Treatment comparison between Placebo and RVT-1401 680 mg/week of Anti-AChR-IgG has been presented

12. Secondary Outcome: Double-Blind Treatment Period: Area Under the Concentration-time Curve From Time 0 to 168 Hours (AUC0-168h) of RVT-1401
Description: Blood samples were collected for the analysis of Pharmacokinetic parameter AUC (0-168h).
Time Frame: Pre-dose; Day 1, Day 3, Day 5, Day 8, Day 15, Day 22, Day 29, Day 36, Day 38, Day 40, Week 7, Week 8
Population: Pharmacokinetic (PK) Analysis Set comprised of all participants who underwent PK sampling and had evaluable concentration-time data for analysis. As PK analyses were not conducted, a PK Analysis Set was not presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 5 | 6
Hours*microgram per milliliter | NA (NA) — Not applicable (NA) indicates data was not available as all concentration values were below the lower limit of quantification. | NA (NA) — NA indicates data was not available as all concentration values were below the lower limit of quantification.

13. Secondary Outcome: Open-label Extension Period: AUC0-168h of RVT-1401
Description: Pharmacokinetic parameters were not estimated because the sparse PK sampling schedule did not allow for accurate estimates of these parameters.
Time Frame: Pre-dose; Day 1, Day 3, Day 5, Day 8, Day 15, Day 22, Day 29, Day 36, Day 38, Day 40, Week 7, Week 8, Week 9, Week 12 and Week 14
Population: Pharmacokinetic Analysis Set. Participants were analyzed based on the randomization schedule, regardless of the treatment actually received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 5 | 4
Hours*microgram per milliliter | NA (NA) — NA indicates data was not available as all concentration values were below the lower limit of quantification. | NA (NA) — NA indicates data was not available as all concentration values were below the lower limit of quantification.

14. Secondary Outcome: Double-Blind Treatment Period: Maximum Concentration (Cmax) of RVT-1401
Description: Blood samples were collected for the analysis of Pharmacokinetic parameter Cmax.
Time Frame: Pre-dose; Day 1, Day 3, Day 5, Day 8, Day 15, Day 22, Day 29, Day 36, Day 38, Day 40, Week 7, Week 8
Population: Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter
Arm/Group | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 5 | 6
micrograms per milliliter | NA (NA) — NA indicates data was not available as all concentration values were below the lower limit of quantification. | NA (NA) — NA indicates data was not available as all concentration values were below the lower limit of quantification.

15. Secondary Outcome: Open-label Extension Period: Cmax of RVT-1401
Description: Blood samples were collected for the analysis of Pharmacokinetic parameter Cmax.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 5 | 4
Micrograms per milliliter | NA (NA) — NA indicates data was not available as all concentration values were below the lower limit of quantification. | NA (NA) — NA indicates data was not available as all concentration values were below the lower limit of quantification.

16. Secondary Outcome: Double-Blind Treatment Period: Trough Concentrations (Ctrough) of RVT-1401
Description: Blood samples were planned to be collected at indicated time points to measure the concentration of RVT-1401 pre-dose (Ctrough) as an assessment of the pharmacokinetic RVT-1401.
Time Frame: Pre-dose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Milligrams per liter
Arm/Group | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 5 | 6
Milligrams per liter | NA (NA) — NA indicates data could not be calculated for double-blind treatment period due to high proportion of non-quantifiable values. | NA (NA) — NA indicates data could not be calculated for double-blind treatment period due to high proportion of non-quantifiable values.

17. Secondary Outcome: Open-label Extension Period: Ctrough of RVT-1401
Description: as for outcome 16
Time Frame: Pre-dose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Milligrams per liter
Arm/Group | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 5 | 4
Milligrams per liter | NA (NA) — NA indicates data could not be calculated for Open-label treatment period due to high proportion of non-quantifiable values. | NA (NA) — NA indicates data could not be calculated for Open-label treatment period due to high proportion of non-quantifiable values.

18. Secondary Outcome: Double-blind Treatment Period: Change From Baseline in the Quantitative Myasthenia Gravis Score (QMG) Score
Description: The QMG score is a physician-reported outcome measure was used to assess MG disease severity and pattern of deficits based on quantitative testing of affected muscle groups. The scale comprised of 13 test items that were graded on a scale of 0 (no myasthenic findings) to 3 (maximal myasthenic deficits). The total sum across all 13 items represents the QMG score. QMG total scores range from 0 to 39 for a given visit, with higher scores indicating more severe disease. Baseline was defined as the last non-missing value prior to the date (time) of first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and at Week 2, Week 3, Week 4, Week 5, Week 6 (Day 36) and Week 7
Population: Full Analysis Set. Only those participants with data available at specified time points has been represented (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 6 | 5 | 6
Scores on a scale
  Week 2, n=6,5,6 | -3.3 (2.16) | -2.8 (5.36) | -1.7 (3.14)
  Week 3, n=6,5,6 | -2.5 (2.74) | -4.6 (7.70) | -2.5 (2.95)
  Week 4, n=6,5,5: number analyzed (Participants) | 6 | 5 | 5
  Week 4, n=6,5,5 | -2.7 (2.73) | -3.6 (6.43) | -3.6 (4.16)
  Week 5, n=6,5,5: number analyzed (Participants) | 6 | 5 | 5
  Week 5, n=6,5,5 | -2.7 (2.73) | -3.2 (6.80) | -3.2 (3.70)
  Week 6 (Day 36), n=6,5,5: number analyzed (Participants) | 6 | 5 | 5
  Week 6 (Day 36), n=6,5,5 | -3.0 (3.22) | -4.0 (6.75) | -4.4 (3.71)
  Week 7, n=5,5,5: number analyzed (Participants) | 5 | 5 | 5
  Week 7, n=5,5,5 | -1.8 (3.27) | -4.0 (6.82) | -3.8 (4.76)

19. Secondary Outcome: Double-Blind Treatment Period: Percentage of Participants With an Improvement/ Response on the QMG Score From Baseline
Description: The response is defined as improvement from Baseline on the QMG score by => 3 points. The QMG score is a physician-reported outcome measure was used to assess MG disease severity and pattern of deficits based on quantitative testing of affected muscle groups. The scale comprised of 13 test items that were graded on a scale of 0 (no myasthenic findings) to 3 (maximal myasthenic deficits). The total sum across all 13 items represents the QMG score. QMG total scores range from 0 to 39 for a given visit, with higher scores indicating more severe disease. Baseline was defined as the last non-missing value prior to the date (time) of first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) to Week 7
Population: Full Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Number; unit: Percentage of participants
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 5 | 5 | 5
Percentage of participants | 20.0 | 40.0 | 60.0

20. Secondary Outcome: Double-Blind Treatment Period: Change From Baseline in the Myasthenia Gravis Activities of Daily Living (MG-ADL) Score
Description: The MG-ADL is an 8-item, participant-reported outcome measure that assessed Myasthenia Gravis symptoms and their effects on activities of daily living, with each response graded from 0 (normal) to 3 (most severe). The MG-ADL score was calculated by totaling the rating for each of the 8 items. Total MG-ADL scores range from 0 to 24 with higher scores indicating more severe disease. Baseline was defined as the last non-missing value prior to the date (time) of first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and at Week 2, Week 3, Week 4, Week 5, Week 6 (Day 36), Week 7
Population: Full Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 6 | 5 | 6
Scores on a scale
  Week 2 | -1.7 (2.34) | -3.2 (6.61) | -0.7 (0.82)
  Week 3 | -0.8 (2.04) | -3.8 (5.97) | -1.7 (1.97)
  Week 4: number analyzed (Participants) | 6 | 5 | 5
  Week 4 | -0.8 (2.64) | -3.2 (6.38) | -2.0 (2.35)
  Week 5: number analyzed (Participants) | 6 | 5 | 5
  Week 5 | -1.5 (3.02) | -3.2 (6.65) | -2.0 (2.35)
  Week 6 (Day 36): number analyzed (Participants) | 6 | 5 | 5
  Week 6 (Day 36) | -1.2 (3.19) | -5.2 (7.09) | -3.4 (3.36)
  Week 7: number analyzed (Participants) | 6 | 5 | 5
  Week 7 | -0.2 (2.71) | -4.4 (7.06) | -3.2 (3.11)

21. Secondary Outcome: Double-Blind Treatment Period: Percentage of Participants With an Improvement/ Response on the MG-ADL Score
Description: The response was defined as improvement (decrease) from Baseline on the MG-ADL score by => 2 points. The MG-ADL is an 8-item, participant-reported outcome measure that assessed Myasthenia Gravis symptoms and their effects on activities of daily living, with each response graded from 0 (normal) to 3 (most severe). The MG-ADL score was calculated by totaling the rating for each of the 8 items. Total MG-ADL scores range from 0 to 24 with higher scores indicating more severe disease. Baseline was defined as the last non-missing value prior to the date (time) of first dose of study drug.
Time Frame: Baseline (Day 1) to Week 7
Population: Full Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Number; unit: Percentage of participants
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 6 | 5 | 5
Percentage of participants | 33.3 | 60.0 | 60.0

22. Secondary Outcome: Double-Blind Treatment Period: Change From Baseline in the Myasthenia Gravis Composite Score (MGC) Score
Description: The MGC was developed by selecting the best performing items from 3 commonly used Myasthenia Gravis specific scales (QMG, Myasthenia Gravis manual muscle test, and MG-ADL) and is comprised of 10 functional domains: 3 ocular, 3 bulbar, 1 respiratory, 1 neck, and 2 limb items. The total score ranges from 0 (no myasthenic findings) to 50 (maximal myasthenic deficits). The scale measures symptoms and signs of MG in these domains incorporating both physician and participant-reported test items. Higher scores correlate with clinical worsening of the disease. Baseline was defined as the last non-missing value prior to the date (time) of first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and at Week 2, Week 3, Week 4, Week 5, Week 6 (Day 36), Week 7
Population: Full Analysis Set. Only those participants with data available at specified timepoints has been presented.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 6 | 5 | 6
Scores on a scale
  Week 2 | -2.3 (2.94) | -7.0 (9.27) | -3.0 (3.10)
  Week 3 | -1.3 (5.20) | -8.8 (9.98) | -2.3 (2.88)
  Week 4: number analyzed (Participants) | 6 | 5 | 5
  Week 4 | -2.0 (8.10) | -7.2 (10.40) | -4.0 (6.60)
  Week 5: number analyzed (Participants) | 6 | 5 | 5
  Week 5 | -4.3 (7.50) | -7.0 (10.07) | -2.8 (4.97)
  Week 6 (Day 36): number analyzed (Participants) | 6 | 5 | 5
  Week 6 (Day 36) | -2.5 (8.04) | -10.4 (9.32) | -6.6 (5.13)
  Week 7: number analyzed (Participants) | 5 | 5 | 5
  Week 7 | -0.8 (7.33) | -9.0 (10.12) | -7.0 (5.34)

23. Secondary Outcome: Double-Blind Treatment Period: Percentage of Participants With an Improvement on the MGC Score
Description: The response was defined as improvement (decrease) from Baseline on the MGC score by => 3 points. The MGC was developed by selecting the best performing items from 3 commonly used Myasthenia Gravis specific scales (QMG, Myasthenia Gravis manual muscle test, and MG-ADL) and is comprised of 10 functional domains: 3 ocular, 3 bulbar, 1 respiratory, 1 neck, and 2 limb items. The total score ranges from 0 (no myasthenic findings) to 50 (maximal myasthenic deficits). The scale measures symptoms and signs of MG in these domains incorporating both physician and participant-reported test items. Higher scores correlate with clinical worsening of the disease. Baseline was defined as the last non-missing value prior to the date (time) of first dose of study drug.
Time Frame: Baseline (Day 1) to Week 7
Population: Full Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Number; unit: Percentage of participants
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 5 | 5 | 5
Percentage of participants | 40.0 | 60.0 | 60.0

24. Secondary Outcome: Double-Blind Treatment Period: Change From Baseline in the Myasthenia Gravis Quality of Life 15 Revised Score (MG-QOL 15r) Score
Description: The MG-QOL15r is a participant-reported questionnaire designed to assess how a participant's Myasthenia Gravis affects different aspects related to their quality of life. The scale includes 15 items that are graded on a scale of 0 to2; the total across is the sum of all 15 items and represents the MG-QOL15r score. The range of the MG-QOL15r score is 0 - 30. Higher scores indicate worse outcomes. Baseline was defined as the last non-missing value prior to the date (time) of first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and at Week 4 and Week 7
Population: Full Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 6 | 5 | 4
Scores on a scale
  Week 4 | -3.5 (3.83) | -6.0 (9.77) | 1.6 (5.03)
  Week 7 | -2.3 (3.93) | -6.6 (10.55) | 2.0 (4.42)

25. Secondary Outcome: Double-Blind Treatment Period: Number of Participants Reporting Confirmed Positive Anti-RVT-1401 Antibodies
Description: The serum levels of anti-RVT-1401 antibodies were determined. All samples that were potentially positive were analyzed with the confirmation assay where presence of anti-RVT-1401 was confirmed; the therapeutic antibody was used to compete with the analytical responses of anti-drug antibody (ADA) to assess specificity of screened positive samples.
Time Frame: Up to Week 7
Population: Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 6 | 5 | 6
Participants | 2 | 1 | 1

26. Secondary Outcome: Open-Label Extension Period: Number of Participants Reporting Confirmed Positive Anti-RVT-1401 Antibodies
Description: The serum levels of anti-RVT-1401 antibodies were determined. All samples that were potentially positive were analyzed with the confirmation assay where presence of anti-RVT-1401 was confirmed; the therapeutic antibody was used to compete with the analytical responses of ADA to assess specificity of screened positive samples.
Time Frame: Up to Week 18
Population: Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week
Number analyzed (Participants) | 6 | 5 | 4
Participants | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline and Up to Week 18
Description: Adverse events and Serious adverse events were collected in Safety Analysis Set in Double-Blind Treatment Period and in OLE Analysis Set in Open-Label Extension Period. Safety Analysis Set comprised of all participants who received at least 1 dose of study medication. OLE Analysis Set comprised of all participants who enrolled in the OLE study phase and received at least 1 dose of study medication in the OLE.
Groups:
- Double-blind Treatment Period: Placebo: Participants were randomized to receive Placebo during the 6-week double blind period. Participants who completed DB Treatment period entered an OLE where they received 340 mg RVT-1401 every 2 weeks (Q2W) x 3 doses, followed by a 6-week follow-up period where the participant did not receive any study treatment. Participants
- Double-blind Treatment Period: RVT-1401 680 mg/Week: Participants were randomized to receive 680 mg/week during the 6-week double blind period. Participants who completed DB Treatment period entered an OLE where they received 340 mg RVT-1401 Q2W x 3 doses, followed by a 6-week follow-up period where the participant did not receive any study treatment. Participants
Arm/Group | Double-blind Treatment Period: Placebo | Double-blind Treatment Period: RVT-1401 340 mg/Week | Double-blind Treatment Period: RVT-1401 680 mg/Week | Open-label Extension Period: RVT-1401 340 mg Biweekly
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/6 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 1/6 | 1/15
Other Adverse Events (participants affected / at risk) | 5/6 | 4/5 | 5/6 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Treatment Period: Placebo (N=6) | Double-blind Treatment Period: RVT-1401 340 mg/Week (N=5) | Double-blind Treatment Period: RVT-1401 680 mg/Week (N=6) | Open-label Extension Period: RVT-1401 340 mg Biweekly (N=15)
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Treatment Period: Placebo (N=6) | Double-blind Treatment Period: RVT-1401 340 mg/Week (N=5) | Double-blind Treatment Period: RVT-1401 680 mg/Week (N=6) | Open-label Extension Period: RVT-1401 340 mg Biweekly (N=15)
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 1 | 2 | 1 | 2
Injection site bruising (General disorders) | 0 | 1 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 1 | 0
Injection site swelling (General disorders) | 1 | 1 | 0 | 1
Vessel puncture site bruise (General disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Red blood cell count increased (Investigations) | 0 | 1 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 1 | 0 | 0
Total complement activity decreased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 3 | 1 | 0 | 2
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT03863080/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT03863080/SAP_001.pdf